CLINICAL TRIAL: NCT04303312
Title: Clinical Evaluation of Solcosreyl and Pumpkin Seed Oil Versus Benzydamine Hydrochloride in Management of Patients With Chemotherapy and Radiotherapy Induced Oral Mucositis
Brief Title: Treatment of Chemotherapy and Radiotherapy Induced Oral Mucositis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ghada zaki (Other)
Responsible Party: Sponsor-Investigator, Ghada zaki, assistant lecturer at el ahram canadian university, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OMED 2_2_1
Record Dates: First submitted 2020-03-04; First posted 2020-03-11 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: Mucositis Oral
Keywords: Oral Mucositis; Pumpkin seed oil; Solcoseryl
MeSH Terms: conditions — Stomatitis | interventions — Benzydamine; Actihaemyl

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant, Care Provider
Masking Description: Treatment will be placed in identical spray containers
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Benzydamine Hydrochloride (Active Comparator): Control Group:Benzydamine Hydrochloride spray by mouth three times daily for 20 days.
  Follow up: The patients will be recalled at one week interval for 20 days.
  Interventions: Combination Product: Solcoseryl and pumpkin seed oil
- 90%solcoseryl and 10% pumpkin seed oil (Experimental): Intervention group: 90% solcoseryl and 10% pumpkin seed oil spray by mouth three times daily for 20 days
  Interventions: Other: Benzydamine Hydrochloride

INTERVENTIONS:
Other: Benzydamine Hydrochloride — Patients will rinse by mouth three times daily for 20 days
  Arms: 90%solcoseryl and 10% pumpkin seed oil
Combination Product: Solcoseryl and pumpkin seed oil — Patients will receive by mouth three times daily for 20 days
  Arms: Benzydamine Hydrochloride

SUMMARY:
Oral mucositis consequences can range from pain, decreased oral intake, impaired speech and swallowing to adverse events as severe as septicemia, increased hospitalization, and G-tube feeding A wide variety of agents have been tested to prevent OM or reduce its severity.This trial will assess the usefulness of solcoseryl and pumpkin seed oil versus Benzydamine Hydrochloride mouth wash in management of oral mucositis in patients receiving radiotherapy and/or chemotherapy.

DETAILED DESCRIPTION:
The term "mucositis" was introduced to describe inflammation of the oral mucosa induced by radiotherapy, chemotherapy and bone marrow transplantation. At present, oral mucositis is considered to be the most serious non-hematological complication of cancer treatment.

Numerous predisposing factors have been blamed for oral mucositis, including: the type of tumor involved, age of the patient, dental health, the nutritional condition of the patient, the maintenance of kidney and liver function and the type of cytostatic agent used.

Clinically, oral Mucositis may appear as erythema, edema or ulceration that can be accompanied by alterations ranging from mild burning sensation to large and painful ulcers that wor¬sen patient's quality of life and limit basic oral functions such as speech, swallowing of saliva or eating.

According to Multinational Association for Supportive Care in cancer and the International Society of Oral Oncology (MASCC/ISOO) guidelines for the management of mucositis, Management of oral mucositis is divided into the following sections: nutritional support, pain control, oral decontamination, palliation of dry mouth, management of oral bleeding and therapeutic interventions for oral mucositis.

Since the primary symptom of oral mucositis is pain which significantly affects nutritional intake, mouth care and quality of life, thus, management of mucositis pain is a primary component of any mucositis management strategy. Use of saline mouth rinses, ice chips and topical mouthrinses containing an anesthetic such as 2% viscous lidocaine can help in reducing pain

Based on the pathogenesis of mucositis with complex biological inflammatory pathways, various therapeutic approach have been proposed to improve oral mucositis.

The current guidelines recommend the use of non-medicated oral rinses such as Benzydamine hydrochloride mouthwash and the use of short term pain killers. Benzydamine hydrochloride - which is a non-steroidal anti-inflammatory drug - can be used in the form of mouth rinse to reduce the severity of oral mucositis. Other management strategies include cryotherapy before the start of chemotheraputic agent administration and application of low-level laser therapy. Palifermin (Keratinocyte growth factor) is the only recommended preventive measure recommended by the ESMO Clinical Practice Guidelines.

Solcoseryl, is a protein free standardized dialysate of calf blood extracted by ultrafiltration. The main constituents of Solcoseryl are inorganic electrolytes (chloride, phosphate, sodium, potassium, calcium, and magnesium) and low-molecular weight substances, including amino acids, biogenic amines and polyamines, sphingolipids, hexoses, eicosanoids, lactate, acetate, succinate, choline, vitamins, adenosine monophosphate (AMP) and inositol phospho-oligosaccharides.

Solcoseryl has a number of beneficial effects. The most important of them include enhanced cellular glucose uptake, improvement of oxygen utilization and energy metabolism , neuroprotective effects, reduction of oxidative stress and apoptosis, accelerated wound healing and improvement of blood microcirculation.

Pumpkin seed oils are good source of vitamins, minerals and anti-oxidants. Active components include fatty acid, 19.4% saturated fatty acids (palmitic acid and stearic acid), 80.7% unsaturated fatty acids (linoleic acid and oleic acid) , Tocopherol (β-tocopherol, γ-tocopherol, δ-tocopherol), carotenoids including β-carotene and lutein, Phytosterols or plant sterols, Amino acid Glutamic and aspartic acid, leucine, valine, phenylalanine, and tryptophan are among the amino acids identified. It has many therapeutic activities like antioxidant activity, anti inflammatory, antimicrobial activity, and anti carcinogenic effect. It is thus a good candidate to counteract the ongoing development of oral mucositis.

ELIGIBILITY:
A- Inclusion criteria:

1. Patients having clinical signs of chemotherapy-induced or radiotherapy-induced OM (WHO oral mucositis grading scale: Grade II, III and IV)
2. Patients over the age of 18 years
3. Patients having no history of allergy, allergic rhinitis and asthma

B- Exclusion criteria:

1. Patients allergic to the used treatment
2. Patient receiving systemic steroids
3. Patients who don't approve to participating in the clinical trial.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Clinical improvement | 20 days
  World Health Organization (WHO)scale.It is graded from 0 to 4. If the patient has no signs and symptoms, it is graded as 0. If the patient has painless ulcers, edema, or mild soreness, it is graded as 1. If there is painful erythema, edema, or ulcers but able to eat, it is graded as 2. If there is painful erythema, edema, or ulcers but unable eat, it is graded as 3. If there a requirement for parenteral or enteral support, it is graded as 4

SECONDARY OUTCOMES:
Quality of life | 20 days
  Patient-Reported Oral Mucositis( PROMS scale) will measure Quality of life .The PROMS scale consists of 10, 100-mm horizontal visual analogue scales addressing oral functions affected by oral mucositis. Participants will be asked to mark a point on the line that best represents their present intra-oral condition.During the baseline examination and prior to their completion of the actual PROMS scale questionnaire, participants were subjected to a few training test-visual analogue scale questions focused on simple everyday topics to familiarize them with the concept of visual analogue scale assisted measurements. The participants will complete the PROMS questionnaire thrice; baseline, after the first week, and at the end of the study after the second week.